CLINICAL TRIAL: NCT04165304
Title: Impact on Drinking Behaviour in Sixth-grade Students Through Changing the School Environment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Since schools are closed due to the current corona virus situation, the study cannot be continued.
Sponsor: Special Institute for Preventive Cardiology And Nutrition (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Version 1.4
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2019-11

CONDITIONS: Students of the 6. Grade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): the range of products offered by the vending machines remains unchanged
- Intervention group 1 (Other): vending machines will be re-equipped to contain 60% drinks containing a maximum of 6.7g sugar/100ml, 20% drinks containing more than 6.7g sugar/100ml and 20% water
  Interventions: Dietary Supplement: sugar reduction
- Intervention group 2 (Other): In the second intervention group, the vending machines offer 80% water and 20% products with a maximum of 6.7g sugar/100ml.
  Interventions: Dietary Supplement: sugar reduction

INTERVENTIONS:
Dietary Supplement: sugar reduction — sugar reduction in the offered drinks
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
This study evaluates the effect of changes in the range of drinks offered in vending machines in schools on the sugar intake of pupils via drinks.

DETAILED DESCRIPTION:
Children and adolescents consume a considerable amount of liquid in the form of sugary drinks. A high sugar diet associated not only with the increase in overweight children, but also with type II diabetes, cardiovascular disease and cancer.

In many schools, cold drink vending machines with different fillings are available offering various sugary drinks.

Participating schools will be randomised in a ratio of 1:1:1 into three groups. In one intervention group, the vending machines will be re-equipped to contain 60% drinks containing a maximum of 6.7g sugar/100ml, 20% drinks containing more than 6.7g sugar/100ml and 20% water. In the second intervention group, the vending machines offer 80% water, 20% products with a maximum of 6.7g sugar/100ml. In the control group, the range of products offered by the vending machines remains unchanged. Information of the students drinking habits, total fluid intake and sugar intake in the form of food and drinks will be collected. In addition, data such as body height, body weight, physical activity and socio-democratic or socio-economic data will be accumulated. The sales figures of the drinks in the vending machines will be recorded and information about the surroundings of the schools (fast food chains, supermarkets, etc.) will be collected.

The survey of students and data collection will be repeated three times. In a sub-study, demographic data and the frequency of consumption of sugared beverages and water are collected from 2 focus groups. In addition, participants will complete a questionnaire on general attitudes towards sugary drinks or water, obstacles to and incentives for reducing sugar consumption by liquids or increasing water consumption.

ELIGIBILITY:
Inclusion Criteria:

* Students in one of the recruited schools
* Appropriate knowledge of the German language

Exclusion Criteria:

* No signed consent of parent and of child

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 431 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Consumption of mean liquid free sugar intake per week (g) by using the 7-day fluid record | 1 week
  self report of fluid consumption

SECONDARY OUTCOMES:
Absolute (mL) and relative (%) contribution of each fluid intake category to total fluid intake by using the 7-day fluid record | 1 week
  self report of fluid consumption, the measure presents only one outcome "fluid intake", which will be reported in "ml" and "%".
Water intake by using the 7-day fluid record with the proportion of children meeting the EFSA adequate intake for water from fluids | 1 week
  self report of fluid consumption
Consumption of free sugar from food by 24-h dietary recall | 24 hours
  self report of food consumption
Body weight and Body-Mass-Index (BMI) by using body weight and height | Start, 3-4 months, 7-8 months
  Measured with a calibrated body scale in light clothes and without shoes
Abdominal girth | Start, 3-4 months, 7-8 months
  inelastic tape
Physical activity | Start, 3-4 months, 7-8 months
  International Physical Activity Questionnaire for Adolescents (IPAQ-A), scale title "Physical activity of adolescents", scale minimum "0", scale maximum "7", higher scores mean a better outcome
Socio-demographic and socioeconomic factors | after 7-8 months
  questionnaire, scale title "socio-demographic and socio-econimoc status", scale minimum is "0", scale maximum is "3", higher scores mean a better outcome
Sales data (frequencies of beverages) of the vending machine and school cafeteria operators | through study completion, an average of 8 month
  Interview

CONTACTS AND LOCATIONS:
Locations (15):
- Austria (15):
  - NMS St. Veit/Glan, Sankt Veit an der Glan, Carinthia
  - NMS II Spittal/Drau, Spittal an der Drau, Carinthia
  - Sport-Mittelschule Matzen-Raggendorf, Matzen, Gänserndorf
  - Gymnasium Bad Vöslau/Gainfard, Bad Vöslau, Lower Austria
  - NMS Lanzenkirchen, Lanzenkirchen, Lower Austria
  - BG/BRG Zehnergasse, Wiener Neustadt, Lower Austria
  - Bischöfliches Gymnasium Graz, Graz, Styria
  - NMS Liezen, Liezen, Styria
  - BG/BRG Wels, Wels, Upper Austria
  - GRG II Zirkusgasse, Vienna
  - BRG Marchettigasse, Vienna
  - GRG Gottschalkgasse, Vienna
  - GWIKU 18 Haizingergasse, Vienna
  - LWS Donaustadt, Vienna
  - GRG 23, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Popkin BM, D'Anci KE, Rosenberg IH. Water, hydration, and health. Nutr Rev. 2010 Aug;68(8):439-58. doi: 10.1111/j.1753-4887.2010.00304.x. PMID 20646222
- [Background] Duffey KJ, Poti J. Modeling the Effect of Replacing Sugar-Sweetened Beverage Consumption with Water on Energy Intake, HBI Score, and Obesity Prevalence. Nutrients. 2016 Jun 28;8(7):395. doi: 10.3390/nu8070395. PMID 27367719
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Background] Han E, Powell LM. Consumption patterns of sugar-sweetened beverages in the United States. J Acad Nutr Diet. 2013 Jan;113(1):43-53. doi: 10.1016/j.jand.2012.09.016. PMID 23260723
- [Background] Luger M, Lafontan M, Bes-Rastrollo M, Winzer E, Yumuk V, Farpour-Lambert N. Sugar-Sweetened Beverages and Weight Gain in Children and Adults: A Systematic Review from 2013 to 2015 and a Comparison with Previous Studies. Obes Facts. 2017;10(6):674-693. doi: 10.1159/000484566. Epub 2017 Dec 14. PMID 29237159
- [Background] Malik VS, Pan A, Willett WC, Hu FB. Sugar-sweetened beverages and weight gain in children and adults: a systematic review and meta-analysis. Am J Clin Nutr. 2013 Oct;98(4):1084-102. doi: 10.3945/ajcn.113.058362. Epub 2013 Aug 21. PMID 23966427
- [Background] Te Morenga L, Mallard S, Mann J. Dietary sugars and body weight: systematic review and meta-analyses of randomised controlled trials and cohort studies. BMJ. 2012 Jan 15;346:e7492. doi: 10.1136/bmj.e7492. PMID 23321486
- [Background] Ma Y, He FJ, Yin Y, Hashem KM, MacGregor GA. Gradual reduction of sugar in soft drinks without substitution as a strategy to reduce overweight, obesity, and type 2 diabetes: a modelling study. Lancet Diabetes Endocrinol. 2016 Feb;4(2):105-14. doi: 10.1016/S2213-8587(15)00477-5. Epub 2016 Jan 7. PMID 26777597
- [Background] Greenwood DC, Threapleton DE, Evans CE, Cleghorn CL, Nykjaer C, Woodhead C, Burley VJ. Association between sugar-sweetened and artificially sweetened soft drinks and type 2 diabetes: systematic review and dose-response meta-analysis of prospective studies. Br J Nutr. 2014 Sep 14;112(5):725-34. doi: 10.1017/S0007114514001329. Epub 2014 Jun 16. PMID 24932880
- [Background] Marshall TA, Levy SM, Broffitt B, Warren JJ, Eichenberger-Gilmore JM, Burns TL, Stumbo PJ. Dental caries and beverage consumption in young children. Pediatrics. 2003 Sep;112(3 Pt 1):e184-91. doi: 10.1542/peds.112.3.e184. PMID 12949310
- [Background] Wilder JR, Kaste LM, Handler A, Chapple-McGruder T, Rankin KM. The association between sugar-sweetened beverages and dental caries among third-grade students in Georgia. J Public Health Dent. 2016 Winter;76(1):76-84. doi: 10.1111/jphd.12116. Epub 2015 Sep 4. PMID 26339945
- [Background] Basu S, McKee M, Galea G, Stuckler D. Relationship of soft drink consumption to global overweight, obesity, and diabetes: a cross-national analysis of 75 countries. Am J Public Health. 2013 Nov;103(11):2071-7. doi: 10.2105/AJPH.2012.300974. Epub 2013 Mar 14. PMID 23488503
- [Background] Singh GM, Micha R, Khatibzadeh S, Shi P, Lim S, Andrews KG, Engell RE, Ezzati M, Mozaffarian D; Global Burden of Diseases Nutrition and Chronic Diseases Expert Group (NutriCoDE). Global, Regional, and National Consumption of Sugar-Sweetened Beverages, Fruit Juices, and Milk: A Systematic Assessment of Beverage Intake in 187 Countries. PLoS One. 2015 Aug 5;10(8):e0124845. doi: 10.1371/journal.pone.0124845. eCollection 2015. PMID 26244332
- [Background] Singh GM, Micha R, Khatibzadeh S, Lim S, Ezzati M, Mozaffarian D; Global Burden of Diseases Nutrition and Chronic Diseases Expert Group (NutriCoDE). Estimated Global, Regional, and National Disease Burdens Related to Sugar-Sweetened Beverage Consumption in 2010. Circulation. 2015 Aug 25;132(8):639-66. doi: 10.1161/CIRCULATIONAHA.114.010636. Epub 2015 Jun 29. PMID 26124185
- [Background] Reichelt AC, Killcross S, Hambly LD, Morris MJ, Westbrook RF. Impact of adolescent sucrose access on cognitive control, recognition memory, and parvalbumin immunoreactivity. Learn Mem. 2015 Mar 16;22(4):215-24. doi: 10.1101/lm.038000.114. Print 2015 Apr. PMID 25776039
- [Background] Yu CJ, Du JC, Chiou HC, Feng CC, Chung MY, Yang W, Chen YS, Chien LC, Hwang B, Chen ML. Sugar-Sweetened Beverage Consumption Is Adversely Associated with Childhood Attention Deficit/Hyperactivity Disorder. Int J Environ Res Public Health. 2016 Jul 4;13(7):678. doi: 10.3390/ijerph13070678. PMID 27384573
- [Background] Mennella JA. Ontogeny of taste preferences: basic biology and implications for health. Am J Clin Nutr. 2014 Mar;99(3):704S-11S. doi: 10.3945/ajcn.113.067694. Epub 2014 Jan 22. PMID 24452237
- [Background] Muckelbauer R, Gortmaker SL, Libuda L, Kersting M, Clausen K, Adelberger B, Muller-Nordhorn J. Changes in water and sugar-containing beverage consumption and body weight outcomes in children. Br J Nutr. 2016 Jun;115(11):2057-66. doi: 10.1017/S0007114516001136. Epub 2016 Apr 4. PMID 27040694
- [Background] Puffer S, Torgerson DJ, Watson J. Cluster randomized controlled trials. J Eval Clin Pract. 2005 Oct;11(5):479-83. doi: 10.1111/j.1365-2753.2005.00568.x. PMID 16164589
- [Background] Ahluwalia N, Dalmasso P, Rasmussen M, Lipsky L, Currie C, Haug E, Kelly C, Damsgaard MT, Due P, Tabak I, Ercan O, Maes L, Aasvee K, Cavallo F. Trends in overweight prevalence among 11-, 13- and 15-year-olds in 25 countries in Europe, Canada and USA from 2002 to 2010. Eur J Public Health. 2015 Apr;25 Suppl 2:28-32. doi: 10.1093/eurpub/ckv016. PMID 25805783
- [Background] Swithers SE, Martin AA, Davidson TL. High-intensity sweeteners and energy balance. Physiol Behav. 2010 Apr 26;100(1):55-62. doi: 10.1016/j.physbeh.2009.12.021. Epub 2010 Jan 6. PMID 20060008
- [Background] Johnson EC, Peronnet F, Jansen LT, Capitan-Jimenez C, Adams JD, Guelinckx I, Jimenez L, Mauromoustakos A, Kavouras SA. Validation Testing Demonstrates Efficacy of a 7-Day Fluid Record to Estimate Daily Water Intake in Adult Men and Women When Compared with Total Body Water Turnover Measurement. J Nutr. 2017 Oct;147(10):2001-2007. doi: 10.3945/jn.117.253377. Epub 2017 Sep 6. PMID 28878034
- [Background] Hagstromer M, Bergman P, De Bourdeaudhuij I, Ortega FB, Ruiz JR, Manios Y, Rey-Lopez JP, Phillipp K, von Berlepsch J, Sjostrom M; HELENA Study Group. Concurrent validity of a modified version of the International Physical Activity Questionnaire (IPAQ-A) in European adolescents: The HELENA Study. Int J Obes (Lond). 2008 Nov;32 Suppl 5:S42-8. doi: 10.1038/ijo.2008.182. PMID 19011653
- [Background] Zhang S, Paul J, Nantha-Aree M, Buckley N, Shahzad U, Cheng J, DeBeer J, Winemaker M, Wismer D, Punthakee D, Avram V, Thabane L. Empirical comparison of four baseline covariate adjustment methods in analysis of continuous outcomes in randomized controlled trials. Clin Epidemiol. 2014 Jul 14;6:227-35. doi: 10.2147/CLEP.S56554. eCollection 2014. PMID 25053894
- [Background] Manachini PL, Parini C, Fortina MG, Benazzi L. BliI, a restriction endonuclease from Bacillus licheniformis. FEBS Lett. 1987 Apr 20;214(2):305-7. doi: 10.1016/0014-5793(87)80075-3. PMID 3032685
- [Background] Grassi E, Evans A, Ranjit N, Pria SD, Messina L. Using a mixed-methods approach to measure impact of a school-based nutrition and media education intervention study on fruit and vegetable intake of Italian children. Public Health Nutr. 2016 Aug;19(11):1952-63. doi: 10.1017/S1368980015003729. Epub 2016 Feb 9. PMID 26857624
- See also: World Health Organization (WHO). Diet, nutrition and the prevention of chronic diseases: report of a Joint WHO/FAO Expert Consultation — https://apps.who.int/iris/bitstream/handle/10665/42665/WHO_TRS_916.pdf;jsessionid=D5FE5BA9BEA21640073612235DFE400D?sequence=1
- See also: Sugars intake for adults and children — https://www.who.int/nutrition/publications/guidelines/sugars_intake/en/
- See also: The Family Affluence Scale as a Measure of National Wealth: Validation of an Adolescent Self-Report Measure — https://link.springer.com/article/10.1007/s11205-005-1607-6